CLINICAL TRIAL: NCT01176487
Title: A Clinical Trial Using 3-Dimensional Conformal Radiation Therapy to Reduce the Toxicity of Palliative Radiation for Lung Cancer
Brief Title: Palliative 3-Dimensional Conformal Radiation Therapy in Reducing Radiation Side Effects in Patients With Lung Cancer. ICORG 06-34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-34 ICORG; ICORG-06-34; EU-21056
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; recurrent small cell lung cancer; extensive stage small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Radiotherapy, Conformal

ARMS (1):
- A (Experimental): A clinical trial using 3-dimensional conformal radiation therapy to reduce the toxicity of palliative radiation for lung cancer
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Radiation: 3-dimensional conformal radiation therapy; Radiation: palliative radiation therapy; Radiation: whole-brain radiation therapy

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy
Radiation: palliative radiation therapy
Radiation: whole-brain radiation therapy

SUMMARY:
RATIONALE: 3-dimensional conformal radiation therapy may lessen side effects caused by palliative radiation therapy and improve the quality of life of patients with lung cancer.

PURPOSE: This clinical trial is studying how well 3-dimensional conformal radiation therapy works in reducing the side effects of palliative radiation in patients with lung cancer.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate that using technically sophisticated 3-dimensional conformal radiation therapy for the palliative treatment of lung cancer patients will result in equivalent degrees of symptom relief and a reduction in the primary endpoint of oesophagitis.

Single arm therapeutic clinical study.

RT Treatment Regimens:

17 Gy/2 fractions or 20Gy/5 fractions or 39Gy/13 fractions

Primary Endpoint:

-The occurrence of Grade 3 or higher oesophagitis in the interval between start and 1-month post completion of treatment as determined by CTCAE Version 4.02

Patients will be assessed pre treatment, during treatment, 2 weeks post completion of treatment, one month post completion of treatment, three months post completion of treatment, and three monthly thereafter

-All patients who complete treatment (and whose on-treatment toxicity is documented) will be evaluable.

Secondary Endpoint:

* Quality of Life Assessment. All patients will be required to complete the EORTC QLQ-C15-PAL (Version 1) and the Lung Specific Module (LC 13)
* The occurrence of other AEs

Safety Endpoint:

-Radio-induced oesophagitis, acute and long term, using the CTCAE Version 4.02.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Karnofsky Performance Status of > or equal to 40%
* Patients with locally advanced or metastatic small cell or non-small cell lung cancer
* The presence of intra-thoracic symptoms requiring palliative treatment
* WBI (if required) is permitted
* The patient's condition must permit waiting for the 3-dimensional design process to be implemented. This will be at the discretion of the Consultant Physician
* Patients presenting with pleural effusions - provided the pleural effusion does not prevent the reasonably accurate delineation of the target volume
* Intra-thoracic disease requiring palliation must be clearly evident on a diagnostic CT scan
* Life expectancy of at least 3 months (assessed by clinician)
* Provision of written informed consent in line with ICH-GCP guidelines

Exclusion Criteria:

-In the opinion of the Investigator, any evidence of severe or uncontrolled systematic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of esophagitis grade 3 or higher according to CTCAE Version 4.02 | 2015
Quality of life as assessed using the EORTC QLQ-C15-PAL (Version 1) questionnaire and the Lung Specific Module (LC 13) | 2015

SECONDARY OUTCOMES:
Local intra-thoracic symptoms | 2015

CONTACTS AND LOCATIONS:
Overall Officials: John Gerard Armstrong, MD, MB, MRCPI, Principal Investigator — Saint Luke's Hospital
Locations (2):
- Ireland (2):
  - St Luke's Radiation Oncology Network (SLRON), Dublin
  - Galway University Hospital, Galway

REFERENCES:
- [Derived] McDermott RL, Armstrong JG, Thirion P, Dunne M, Finn M, Small C, Byrne M, O'Shea C, O'Sullivan L, Shannon A, Kelly E, Hacking DJ. Cancer Trials Ireland (ICORG) 06-34: A multi-centre clinical trial using three-dimensional conformal radiation therapy to reduce the toxicity of palliative radiation for lung cancer. Radiother Oncol. 2018 May;127(2):253-258. doi: 10.1016/j.radonc.2018.02.028. Epub 2018 Mar 13. PMID 29548561